CLINICAL TRIAL: NCT00529542
Title: A Six-week Double Blinded, Randomized Trial of Atorvastatin for the Treatment of PCOS Women With Elevated LDL Cholesterol
Brief Title: A Trial of Lipitor (Atorvastatin) for the Treatment of Polycystic Ovary Syndrome (PCOS) in Women With Elevated Low-density Lipoprotein (LDL) Cholesterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19286
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Atorvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental)
  Interventions: Drug: Lipitor
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lipitor — 40mg caplets per day for six weeks
  Other Names: Atorvastatin
  Arms: Atorvastatin
Drug: Placebo — 1 placebo caplet per day for six weeks.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of Lipitor (Atorvastatin) for the treatment of PCOS with elevated LDL cholesterol.

DETAILED DESCRIPTION:
The investigators hypothesize that improving the lipid profile with atorvastatin will improve vascular function, increase the frequency of ovulation, decrease androgen levels, improve insulin sensitivity, and improve the lipid profile more efficiently than placebo.

ELIGIBILITY:
Inclusion Criteria: Women with PCOS

* 8 or fewer menstrual periods per year
* elevated serum total testosterone
* elevated LDL cholesterol

Exclusion Criteria:

* current pregnancy or breastfeeding
* current use of oral contraceptives, progestins
* insulin sensitizing medications
* thyroid disease, hyperprolactinemia, active liver disease, type 1 or type 2 diabetes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S Hershey Medical Center, College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Xiong T, Fraison E, Kolibianaki E, Costello MF, Venetis C, Kostova EB. Statins for women with polycystic ovary syndrome not actively trying to conceive. Cochrane Database Syst Rev. 2023 Jul 18;7(7):CD008565. doi: 10.1002/14651858.CD008565.pub3. PMID 37462232
- [Derived] Raja-Khan N, Kunselman AR, Hogeman CS, Stetter CM, Demers LM, Legro RS. Effects of atorvastatin on vascular function, inflammation, and androgens in women with polycystic ovary syndrome: a double-blind, randomized, placebo-controlled trial. Fertil Steril. 2011 Apr;95(5):1849-52. doi: 10.1016/j.fertnstert.2010.11.040. Epub 2010 Dec 8. PMID 21144505
- See also: Related Info — http://www.pennstatehershey.org/web/obgyn/research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the clinics of the Departments of Medicine and Obstetrics and Gynecology at Penn State Hershey Medical Center from October 20, 2006 to September 8, 2008.
Groups:
- Atorvastatin: Atorvastatin, 40 mg qd
- Placebo: Placebo qd
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 9 | 11
Completed | 8 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-mediated Dilation (FMD)
Description: Brachial artery FMD, the percent change in brachial artery diameter following release of transient occlusion, was selected as the primary outcome because it is the most widely used research tool for evaluating the effects of interventions on endothelial function. FMD has been shown to predict longterm cardiovascular events, even in patients with no apparent heart disease.
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: % change in brachial artery diameter
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
% change in brachial artery diameter
  Before treatment | 12.0 (7.3) | 9.8 (5.8)
  After treatment | 10.4 (4.6) | 10.2 (2.9)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; This study was initiated as a pilot study with the goal of enrolling 19 women in each group, which we hypothesized would provide 80% power to detect an absolute difference in the change in FMD from baseline between the two groups (Atorvastatin vs. Placebo) of 3.75%, assuming a common standard deviation (SD) of 4%, using a two-sided, two-sample t-test with α=0.05. Recruitment was slow due to strict inclusion/ exclusion criteria so we analyzed our data after the first 20 women completed the study; Test type: Superiority or Other; p = 0.58, Linear mixed-effects models — All hypotheses tests were two-sided; Linear mixed-effects models were fit to continuous outcomes to assess the change from baseline to 6 weeks between groups; Mean Difference (Net) = -2.0, 95% CI 2-sided [-9.3 to 5.3] — This analysis revealed that the required sample size was 235 subjects per group for 80% power to detect an absolute 2% increase in FMD with Atorvastatin vs. Placebo. We stopped the trial because we had insufficient funds for the required sample size

2. Secondary Outcome: Peak Brachial Artery Conductance (BAC)
Description: Pneumatic cuffs were positioned on the upper arm and wrist of the experimental arm. The brachial artery was imaged using an ATL Doppler ultrasound probe (5-12MHz linear array scanhead, HDI 5000, Advanced Technology Laboratories, Bothell, WA). Mean blood flow velocity (MBV) and brachial artery diameter (BAD) were recorded at baseline. Then the wrist cuff was inflated to 200-250 mmHg. After a minute, with the wrist cuff still inflated, the arm cuff was inflated to 200-250 mmHg. After 10 minutes the arm cuff was released to induce reactive hyperemia in the brachial artery. Upon release of the arm cuff, we continuously measured blood pressure (BP), heart rate (HR), and MBV, and intermittently measured BAD in the experimental arm. Brachial artery conductance (BAC)was calculated as MBV/MAP and FMD was calculated as percent change in BAD from baseline.
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: ml/sec/mm Hg
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
ml/sec/mm Hg
  Before treatment | 5.4 (2.9) | 3.6 (3.0)
  After treatment | 6.9 (2.8) | 4.3 (3.3)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; What is being compared for this analysis is the change from baseline for "Atorvastatin" to the change from baseline for "Placebo."; Test type: Superiority or Other; p = 0.39, Linear mixed-effects models; Mean Difference (Net) = 0.7, 95% CI 2-sided [-0.9 to 2.3]

3. Secondary Outcome: Total Cholesterol
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mg/dl
  Before treatment | 215.8 (39.0) | 202.8 (28.3)
  After treatment | 132.0 (19.7) | 192.1 (33.6)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Linear mixed-effects models; Mean Difference (Net) = -70.8, 95% CI 2-sided [-95.2 to -46.4]

4. Secondary Outcome: LDL Cholesterol
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mg/dl
  Before treatment | 140.7 (24.6) | 131.3 (21.6)
  After treatment | 68.5 (19.3) | 118.8 (26.8)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Linear mixed-effects models; Mean Difference (Net) = -57.6, 95% CI 2-sided [-79.3 to -35.9]

5. Secondary Outcome: HDL Cholesterol
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mg/dl
  Before treatment | 44.4 (14.6) | 46.5 (8.6)
  After treatment | 47.8 (11.8) | 46.8 (8.4)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.26, Linear mixed-effects models; Mean Difference (Net) = 3.4, 95% CI 2-sided [-2.7 to 9.5]

6. Secondary Outcome: Triglycerides
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mg/dl
  Before treatment | 153.3 (84.9) | 125.5 (54.2)
  After treatment | 78.5 (24.8) | 132.5 (45.7)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Linear mixed-effects models; Mean Difference (Net) = -82.2, 95% CI 2-sided [-126.2 to -38.1]

7. Secondary Outcome: Fasting Glucose
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mg/dl
  Before treatment | 87.7 (9.0) | 85.3 (8.0)
  After treatment | 87.8 (8.5) | 88.9 (10.7)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.45, Linear mixed-effects models; Mean Difference (Net) = -3.3, 95% CI 2-sided [-12.4 to 5.8]

8. Secondary Outcome: Fasting Insulin
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: uU/ml
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
uU/ml
  Before treatment | 18.6 (10.1) | 16.8 (9.5)
  After treatment | 21.0 (11.8) | 15.9 (6.7)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.33, Linear mixed-effects models; Mean Difference (Net) = 2.5, 95% CI 2-sided [-2.8 to 7.9]

9. Secondary Outcome: Area Under the Curve (AUC) for Glucose During OGTT
Description: A 75 gram oral glucose tolerance test (OGTT) was performed with blood draws at 0, 30, 60, 90 and 120 minutes.
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mg*minute/dL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mg*minute/dL
  Before treatment | 15693 (2162) | 15309 (3692)
  After treatment | 16136 (2569) | 15448 (3165)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.61, Linear mixed-effects models; Mean Difference (Net) = 586, 95% CI 2-sided [-1811 to 2983]

10. Secondary Outcome: AUC for Insulin
Description: Area under the curve for insulin during OGTT: A 75 gram oral glucose tolerance test was performed with blood draws at 0, 30, 60, 90 and 120 minutes.
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: uU*minute/mL
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
uU*minute/mL
  Before treatment | 12738 (10010) | 9338 (5208)
  After treatment | 17479 (11929) | 9132 (4466)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.07, Linear mixed-effects models; Mean Difference (Net) = 3385, 95% CI 2-sided [-287 to 7056]

11. Secondary Outcome: Total Testosterone
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
ng/dl
  Before treatment | 61.3 (16.9) | 92.3 (49.8)
  After treatment | 47.1 (21.4) | 75.7 (43.6)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.88, Linear mixed-effects models; Mean Difference (Net) = 1.8, 95% CI 2-sided [-24.1 to 27.8]

12. Secondary Outcome: Androstenedione
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
ng/ml
  Before treatment | 3.4 (0.8) | 3.8 (1.2)
  After treatment | 2.5 (0.9) | 4.1 (1.2)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Linear mixed-effects models; Mean Difference (Net) = -1.1, 95% CI 2-sided [-1.6 to -0.5]

13. Secondary Outcome: DHEAS
Description: Dehydroepiandrosterone sulfate
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
ng/ml
  Before treatment | 1630.0 (873.1) | 1701.5 (681.3)
  After treatment | 1326.4 (854.3) | 1739.5 (781.8)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.02, Linear mixed-effects models; Mean Difference (Net) = -364.3, 95% CI 2-sided [-655.3 to -73.2]

14. Other Pre Specified Outcome: High-sensitivity C-reactive Protein (hsCRP)
Description: high sensitive C-reactive protein as a measure of inflammation
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mg/L
  Before treatment | 8.0 (9.6) | 7.2 (7.7)
  After treatment | 4.3 (5.4) | 6.0 (7.3)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.21, Linear mixed-effects models; Mean Difference (Net) = -2.4, 95% CI 2-sided [-6.4 to 1.5]

15. Post Hoc Outcome: Systolic Blood Pressure
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mm Hg
  Before treatment | 119.8 (15.8) | 114.5 (14.4)
  After treatment | 112.0 (13.2) | 111.4 (8.8)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.27, Linear mixed-effects models; Mean Difference (Net) = -5.9, 95% CI 2-sided [-16.9 to 5.0]

16. Post Hoc Outcome: Diastolic Blood Pressure
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mm Hg
  Before treatment | 70.8 (14.8) | 64.6 (8.0)
  After treatment | 64.3 (12.3) | 65.4 (8.1)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.05, Linear mixed-effects models; Mean Difference (Net) = -7.8, 95% CI 2-sided [-15.8 to 0.1]

17. Post Hoc Outcome: Mean Ovarian Volume
Description: Pelvic ultrasound was performed using the 6.5 megahertz (MHz) probe of an ATL 400 machine to characterize ovarian size and morphology. Since in vitro studies demonstrate that statins inhibit ovarian theca-interstitial cell proliferation, we hypothesized that statins might reduce ovarian volume in PCOS.
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
mm3
  Before treatment | 15.1 (8.8) | 25.4 (13.7)
  After treatment | 19.2 (7.0) | 25.2 (9.9)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.48, Linear mixed-effects models; Mean Difference (Net) = 3.5, 95% CI 2-sided [-6.8 to 13.7]

18. Post Hoc Outcome: Body Mass Index
Time Frame: baseline and 6 weeks
Population: All analyses were performed by intention-to-treat.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 9 | 11
kg/m2
  Before treatment | 40.1 (11.8) | 36.0 (10.4)
  After treatment | 38.2 (8.4) | 35.8 (10.8)
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.63, Linear mixed-effects models; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.6 to 1.0]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/11
Other Adverse Events (participants affected / at risk) | 1/9 | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=9) | Placebo (N=11)
gallbladder removal (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=9) | Placebo (N=11)
swelling (General disorders) | 0 (0) | 1 (1)
muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No